CLINICAL TRIAL: NCT00176397
Title: PCI With DES Versus CABG for Patients With Significant Left Main Stenosis
Brief Title: Percutaneous Coronary Intervention (PCI) With Drug-Eluting Stents (DES) Versus Coronary Artery Bypass Graft (CABG) for Patients With Significant Left Main Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118/2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Stenosis; Coronary Artery Disease
Keywords: left main coronary artery; coronary artery disease
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (left main)

SUMMARY:
Recent technical advances in percutaneous coronary interventions have made it possible to approach patients with coronary lesions formerly considered to be classical candidates for bypass surgery, e.g. patients with left main coronary stenosis. However, it is still unclear whether the good long-term results achieved with the surgical therapy can be reproduced by an interventional strategy using drug-eluting stents (DES).

The aim of the current trial is, therefore, to compare the clinical and angiographic results of PCI and CABG in patients with left main coronary stenosis.

DETAILED DESCRIPTION:
Recent technical advances in percutaneous coronary interventions have made it possible to approach patients with coronary lesions formerly considered to be classical candidates for bypass surgery, e.g. patients with left main coronary stenosis. However, it is still unclear whether the good long-term results achieved with the surgical therapy can be reproduced by an interventional strategy using drug-eluting stents (DES).

The aim of the current trial is, therefore, to compare the clinical and angiographic results of PCI and CABG in patients with left main coronary stenosis.

The study was planned as a "non-inferiority" trial based on the hypothesis that PCI may be able to reach similar long-term results as compared to CABG.

ELIGIBILITY:
Inclusion Criteria:

* Significant left main coronary stenosis >= 50%

Exclusion Criteria:

* Acute myocardial infarction (STEMI < 48h)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-08

PRIMARY OUTCOMES:
Major adverse coronary events (cardiac death, myocardial infarction, need for repeat revascularisation)

SECONDARY OUTCOMES:
Functional status (CCS-class)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, MD, Study Director — University of Leipzig; Friedrich Mohr, MD, Study Director — University of Leipzig
Locations (1):
- University of Leipzig, Heart Center, Leipzig, Saxony, Germany